CLINICAL TRIAL: NCT01998126
Title: Evaluation of Combination Checkpoint Inhibitor Plus Targeted Inhibitor (Erlotinib or Crizotinib) for EGFR or ALK Mutated Stage IV Non-small Cell Lung Cancer: Phase Ib With Expansion Cohorts
Brief Title: Combination Checkpoint Inhibitor Plus Erlotinib or Crizotinib for EGFR or ALK Mutated Stage IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI66705
Record Dates: First submitted 2013-07-11; First posted 2013-11-28 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ipilimumab; Erlotinib Hydrochloride; Crizotinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- EGFR patients with ipilimumab (Experimental): ipilimumab and erlotinib in EGFR mutated patients
  Interventions: Drug: Ipilimumab; Drug: Erlotinib
- ALK patients plus ipilimumab (Experimental): ipilimumab and crizotinib in ALK mutated patients
  Interventions: Drug: Ipilimumab; Drug: Crizotinib
- EGFR patients with nivolumab (Experimental): nivolumab and erlotinib in EGFR mutated patients
  Interventions: Drug: Erlotinib; Drug: Nivolumab
- ALK patients plus nivolumab (Experimental): nivolumab and crizotinib in ALK mutated patients
  Interventions: Drug: Crizotinib; Drug: Nivolumab

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab 3 mg/kg x 4 (given with standard Erlotinib or Crizotinib based on mutation)
  Other Names: Yervoy
  Arms: ALK patients plus ipilimumab; EGFR patients with ipilimumab
Drug: Erlotinib — Erlotinib 150 mg once daily or current tolerable dose (given with Ipilimumab)
  Arms: EGFR patients with ipilimumab; EGFR patients with nivolumab
Drug: Crizotinib — Crizotinib 250 mg twice daily or current tolerable dose (given with Ipilimumab)
  Arms: ALK patients plus ipilimumab; ALK patients plus nivolumab
Drug: Nivolumab
  Other Names: Nivolumab 240 mg every 2 weeks
  Arms: ALK patients plus nivolumab; EGFR patients with nivolumab

SUMMARY:
The goals of the overall study are to evaluate a recommended phase 2 dose and the short and long term toxicities of the combinations. This is a modified phase I trial of immune checkpoint inhibitors in combination with mutation - specific targeted therapy (crizotinib or erlotinib) at conventional doses stratified for presence of ALK (Anaplastic lymphoma kinase) or EGFR (epidermal growth factor receptor) mutation.

The goals of the overall study are to evaluate a recommended phase 2 dose and the short and long term toxicities of the combinations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Stage IV Non-Small Cell Lung Cancer (NSCLC), or Stages II - III NSCLC that cannot be treated curatively with standard techniques.
* Non-Small Cell Lung Cancer (NSCLC) that is either EGFR or ALK mutated.
* Untreated with/or actively treated with specific inhibitor for less than 6 months if not progressing on active therapy.
* Age > 18.
* ECOG performance status 0, 1 or 2.
* Prior chemotherapy is allowed if > one month from the end of treatment. Patients must not have received chemotherapy within 4 weeks of the start of study drug.
* Brain metastases are allowed if the patient is asymptomatic or previous steroid treatment was discontinued > 6 weeks.
* Adequate bone marrow function as defined in the protocol
* Serum bilirubin levels < 1.5 mg/dL except for patients with Gilbert's syndrome.
* Adequate organ function as defined in the protocol
* If female and of childbearing potential, documentation of negative pregnancy test (serum or urine) within 7 days prior to first dose.
* Able to provide informed consent and have signed an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Concurrent therapy with any other non-protocol anti-cancer therapy.
* History of any other malignancy requiring active treatment.
* Patients who have had a history of acute diverticulitis, intra-abdominal abscess, Gastrointestical obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation.
* History of symptomatic autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre Syndrome). History of vitiligo and adequately controlled endocrine deficiencies such as hypothyroidism are allowed.
* Significant cardiovascular disease including:
* Active, clinically symptomatic left ventricular failure.
* Uncontrolled symptomatic hypertension that cannot be controlled with anti-hypertensive agents.
* Myocardial infarction, severe angina, or unstable angina within 6 months prior to administration of first dose of study drug.
* History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation)
* Cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with anti-arrhythmic medication)
* Coronary or peripheral artery bypass graft within 6 months of screening.
* Uncontrolled CNS metastases are not allowed; subjects with previously treated brain metastases will be allowed if the brain metastases have been treated, toxicities have resolved to grade 1 or baseline and steroids are no longer required. Leptomeningeal metastases are not allowed.
* Serious/active infection or infection requiring parenteral antibiotics.
* Pregnant or lactating females.
* HIV infection or chronic hepatitis B or C. Negative Screening tests for HIV, Hepatitis B, and Hepatitis C are required.
* The presence of any other medical or psychiatric disorder that, in the opinion of the treating physician, would contraindicate the use of the drugs in this protocol or place the subject at undue risk for treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-12-02 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
toxicity of ipilimumab and erlotinib in EGFR mutated patients | 36 months
  The immune-related response criteria (irRC) incorporate several elements reflecting the complex tumor dynamics of ipilimumab/nivolumab treatment. Under these criteria, a measure of tumor volume is used that incorporates the contribution of new measurable lesions. Each net percentage change in tumor burden per assessment using irRC accounts for the size and growth kinetics of both old and new lesions as they appear. New lesions alone do not qualify as immune-related progressive disease.
toxicity of ipilimumab and crizotinib in ALK mutated patients | 36 months
  The immune-related response criteria (irRC) incorporate several elements reflecting the complex tumor dynamics of ipilimumab/nivolumab treatment. Under these criteria, a measure of tumor volume is used that incorporates the contribution of new measurable lesions. Each net percentage change in tumor burden per assessment using irRC accounts for the size and growth kinetics of both old and new lesions as they appear. New lesions alone do not qualify as immune-related progressive disease.
toxicity of nivolumab and erlotinib in EGFR mutated patients | 36 months
  The immune-related response criteria (irRC) incorporate several elements reflecting the complex tumor dynamics of ipilimumab/nivolumab treatment. Under these criteria, a measure of tumor volume is used that incorporates the contribution of new measurable lesions. Each net percentage change in tumor burden per assessment using irRC accounts for the size and growth kinetics of both old and new lesions as they appear. New lesions alone do not qualify as immune-related progressive disease.
toxicity of nivolumab and crizotinib in ALK mutated patients | 36 months
  The immune-related response criteria (irRC) incorporate several elements reflecting the complex tumor dynamics of ipilimumab/nivolumab treatment. Under these criteria, a measure of tumor volume is used that incorporates the contribution of new measurable lesions. Each net percentage change in tumor burden per assessment using irRC accounts for the size and growth kinetics of both old and new lesions as they appear. New lesions alone do not qualify as immune-related progressive disease.

SECONDARY OUTCOMES:
Response rate | 36 months
Progression Free Survival (PFS) | 36 months
Overall Survival | 36 months
immune function pre and post immune therapy | 36 months
  The immune-related response criteria (irRC) incorporate several elements reflecting the complex tumor dynamics of ipilimumab treatment. Under these criteria, a measure of tumor volume is used that incorporates the contribution of new measurable lesions. Each net percentage change in tumor burden per assessment using irRC accounts for the size and growth kinetics of both old and new lesions as they appear. New lesions alone do not qualify as immune-related progressive disease.
  In this study, immune-related response criteria (irRC) will be used to assess subject response to study treatment per investigator assessment. The secondary endpoint irPFS will be determined based on investigator assessment. In order to adequately address this secondary objective, investigators will follow the clinical practice guidelines to obtain additional tumor assessments beyond mWHO PD and follow the instructions in this section for the determination of immune-related response.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Chalmers AW, Patel S, Boucher K, Cannon L, Esplin M, Luckart J, Graves N, Van Duren T, Akerley W. Phase I Trial of Targeted EGFR or ALK Therapy with Ipilimumab in Metastatic NSCLC with Long-Term Follow-Up. Target Oncol. 2019 Aug;14(4):417-421. doi: 10.1007/s11523-019-00658-0. PMID 31346927